CLINICAL TRIAL: NCT03521115
Title: Web-based Family Prevention of Alcohol and Risky Sex for Older Teens
Brief Title: Family Based Prevention of Alcohol and Risky Sex for Older Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: Klein Buendel, Inc. (Industry); University of New Mexico (Other)
Responsible Party: Principal Investigator, Brenda Miller, Senior Scientist, Pacific Institute for Research and Evaluation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AA020977
Record Dates: First submitted 2018-04-16; First posted 2018-05-11 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Alcohol Drinking; Alcohol Intoxication; Alcohol Poison; Alcohol-Related Disorders; Alcohol Impairment; Alcohol Withdrawal; Alcohol Abstinence; Alcohol; Harmful Use; Sex Behavior; Sexual Aggression; Sexual Harassment; Relation, Interpersonal
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication; Alcohol-Related Disorders; Alcohol Abstinence; Sexual Behavior; Sexual Harassment

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: Parents and Teens were either assigned to the full intervention or provided with didactic materials available on the internet. Family is considered the level of participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Choices 4 Teens (Experimental): A web-based intervention consisting of 3 main components (Communication, Alcohol, Relationships) provided to both parents and teens was completed by parents and teens individually. At the end of each component, discussion guidelines were given to promote communications and to offer skill building practices between parent and teen regarding the component topic. Both the parent and teen were required to complete the component and discussion before moving to the next component. Numbers are provided for the number of families
  Interventions: Behavioral: Smart Choices 4 Teens
- Control condition (No Intervention): This group was provided with websites where information was available regarding the same topics.

INTERVENTIONS:
Behavioral: Smart Choices 4 Teens — This is a web-based prevention program designed to convey information about alcohol and relationships and the types of choices that they are making regarding these topics. General communications was another core element of the program that provided parents and teens with some key elements of talking to each other.
  Arms: Smart Choices 4 Teens

SUMMARY:
An online, interactive web-based program for older teens and their parents is designed to address teen alcohol use and teen relationships. The parent-teen dyad both participate in the web-based program and engage in off-line discussion activities. This intervention promotes communication skills, refusal skills, and helps teens consider how to make healthy choices. A total of 411 family dyads (one parent, one teen) were recruited.

DETAILED DESCRIPTION:
This purpose of this study is to develop an interactive, web-based prevention program for parents and older teens that focuses on teen use of alcohol and teen relationships. The study is designed as a randomized controlled trial.

Specific Aim 1: To adapt two parent-based prevention strategies (Family Matters and Parent Handbook) to provide a family-based approach for addressing older teen alcohol related risk behaviors and sexual risk behaviors and sex in combination with alcohol use (hereafter called alcohol and/or sexual risk behaviors) using the web as the program delivery mode.

Specific Aim 2: To test whether exposure to the program leads to expected changes in targeted teen beliefs and behaviors, including reductions in alcohol and/or sexual risk behaviors.

Specific Aim 3: To examine whether program effects on teen alcohol and/or sexual risk behaviors are mediated through changes in intermediate program targeted beliefs (parents and teen) and behaviors (e.g., parent-teen--communication). Program fidelity and process measures may also mediate these outcomes.

Phase I integrates and adapts the two parent-based approaches and creates a web-based interactive delivery of materials. Expert panels, focus groups, and usability assessments will inform the process. Phase II is an RCT with 400 families with the web-based intervention. Surveys will be conducted at baseline, and for three follow-up periods (6, 12, & 18 months). Analyses will examine teen outcomes related to alcohol and/or sexual risk behaviors. Changes in mediators directly impacted by the program for both teens and parents will be examined. Process and fidelity information will be collected and assessed.

A web-based prevention strategy supporting parents and teens, is significant and timely. Parents and teens will use the internet to make health decisions. This program is uniquely different from other programs be-cause it addresses teens at high risk for alcohol and/or sexual risk behaviors. Further, the strategy involves both parents and teens through an interactive framework. The approach utilizes the strengths of Family Matters which promotes specific exercises and activities between parents and teens and the strengths of the Parent Handbook which addresses issues of importance to this age range.

ELIGIBILITY:
Inclusion Criteria:

* One parent and the teen both had to enroll in the study.

Exclusion Criteria:

* Non-English speaking

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 411 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2017-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda A Miller, Ph.D., Principal Investigator — Pacific Institute for Research & Evaluation
Locations (1):
- Brenda Miller, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Byrnes HF, Miller BA, Grube JW, Bourdeau B, Buller DB, Wang-Schweig M, Woodall WG. Prevention of alcohol use in older teens: A randomized trial of an online family prevention program. Psychol Addict Behav. 2019 Feb;33(1):1-14. doi: 10.1037/adb0000442. Epub 2019 Jan 14. PMID 30640504
- [Result] Wang-Schweig M, Miller BA, Buller DB, Byrnes HF, Bourdeau B, Rogers V. Using Panel Vendors for Recruitment Into a Web-Based Family Prevention Program: Methodological Considerations. Eval Health Prof. 2017 Jan 1:163278717742189. doi: 10.1177/0163278717742189. Online ahead of print. PMID 29172702
- [Result] Bourdeau B, Miller BA, Byrnes HF, Woodall WG, Buller DB, Grube JW. Efficacy of a Web-Based Intervention (Smart Choices 4 Teens) for Facilitating Parent-Adolescent Communication About Relationships and Sexuality: Randomized Controlled Trial. JMIR Pediatr Parent. 2021 Jun 15;4(2):e19114. doi: 10.2196/19114. PMID 34128818
- See also: Efficacy of a Web-Based Intervention (Smart Choices 4 Teens) for Facilitating Parent-Adolescent Communication About Relationships and Sexuality: Randomized Controlled Trial — https://pediatrics.jmir.org/2021/2/e19114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2014-November 2015 Recruited national sample from two panel vendors
Pre-assignment Details: To be eligible, one teen and one parent had to be willing to participate. Enrollment was considered complete after the participants completed consent and baseline surveys. A total of 559 families were eligible and 148 of eligible families declined to participate, leaving a total of 411 families.
Groups:
- Smart Choices 4 Teens: A web-based intervention consisting of 3 main components (Communication, Alcohol, Relationships) provided to both parents and teens was completed by parents and teens individually. At the end of each component, discussion guidelines were given to promote communications and to offer skill building practices between parent and teen regarding the component topic. Both the parent and teen were required to complete the component and discussion before moving to the next component.
  Smart Choices 4 Teens: This is a web-based prevention program designed to convey information about alcohol and relationships and the types of choices that they are making regarding these topics. General communications was another core element of the program that provided parents and teens with some key elements of talking to each other.
Period: Time 0 Baseline Surveys
Arm/Group | Smart Choices 4 Teens | Control Condition
Started | 206 | 205
Completed | 206 | 205
Not Completed | 0 | 0
Period: Time 1 Survey (6 Months Post Baseline)
Arm/Group | Smart Choices 4 Teens | Control Condition
Started (Failure to complete program did not preclude completing surveys.) | 206 | 205
Completed | 150 | 165
Not Completed | 56 | 40
Not completed — Lost to Follow-up | 56 | 40
Period: Time 2 Survey (12 Months Post Baseline)
Arm/Group | Smart Choices 4 Teens | Control Condition
Started | 150 | 165
Completed | 147 | 164
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1
Period: Time 3 Survey (18 Months Post Baseline)
Arm/Group | Smart Choices 4 Teens | Control Condition
Started | 147 | 164
Completed | 145 | 164
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smart Choices 4 Teens | Control Condition | Total
Number analyzed (Participants) | 206 | 205 | 411
Age, Continuous [Mean (Standard Deviation); unit: years] — parent and teen ages Population: There are two distinct groups in this study: parents and teens. To show the ages for each group, separate rows have been established
  years
    parent age | 43.73 (7.039) | 43.75 (6.385) | 43.74 (6.711)
    teen age | 16.40 (.492) | 16.34 (.474) | 16.37 (.483)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There is one teen in each group for whom sex is unknown or not specified
  Participants
    Parent Gender: Female | 173 | 175 | 348
    Parent Gender: Male | 33 | 30 | 63
    Teen Gender: number analyzed (Participants) | 205 | 204 | 409
    Teen Gender: Female | 109 | 117 | 226
    Teen Gender: Male | 96 | 87 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Parent Ethnicity: Hispanic or Latino | 16 | 14 | 30
  Parent Ethnicity: Not Hispanic or Latino | 190 | 190 | 380
  Parent Ethnicity: Unknown or Not Reported | 0 | 1 | 1
  Teen Ethnicity: Hispanic or Latino | 21 | 14 | 35
  Teen Ethnicity: Not Hispanic or Latino | 179 | 190 | 369
  Teen Ethnicity: Unknown or Not Reported | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 24 | 24 | 48
  White | 161 | 157 | 318
  More than one race | 13 | 11 | 24
  Unknown or Not Reported | 2 | 7 | 9
Region of Enrollment [Number; unit: participants] — Nationwide sample to reflect diversity of national population
  participants
    United States | 206 | 205 | 411
Any Alcohol Use [Count of Participants; unit: Participants] — Have you had a drink of alcohol in the past 6 months? (A drink is a glass of wine, a can of beer, a wine cooler, a shot glass of liquor, or a mixed drink).(Response category-1=yes and 0=no) Population: Missing data accounts for discrepancy
  Participants
    number analyzed (Participants) | 200 | 198 | 398
    (all) | 21 | 26 | 47
Frequency of Alcohol Use [Mean (Standard Deviation); unit: units on a scale] — Over the past 30 days, how many times have you had a drink of alcohol? (response categories: 0=none, 1=once, 2=2-3 times, 3= once a week, 4=2-3 times a week--higher score is more frequent drinking during the past 30 days) Population: Missing data accounts for discrepancy
  units on a scale
    number analyzed (Participants) | 198 | 200 | 398
    (all) | .21 (.59) | .17 (.54) | .19 (.57)
Quantity of alcohol consumed on drinking days [Mean (Standard Deviation); unit: units on a scale] — Over the past 30 days, how many drinks did you usually have on days you drank? (response categories: 0= less than one, 1, 2, 3, 4, 5, 6, 7= more than six) Population: Missing data accounts for differences in numbers
  units on a scale
    number analyzed (Participants) | 198 | 200 | 398
    (all) | .27 (.93) | .26 (1.05) | .27 (.99)
Number of times drunk or very, very high [Mean (Standard Deviation); unit: units on a scale] — Over the past 6 months, how many times have you gotten drunk or very, very high on alcohol? (Response categories: 0=none, 1=once a month, 2=2-3 times a month, 3=once a week, 4= 2-3 times a week, 5=daily or almost daily). Population: Missing data accounts for discrepancy
  units on a scale
    number analyzed (Participants) | 200 | 200 | 400
    (all) | .29 (.89) | .24 (.74) | .26 (.82)
Parental approval of teen drinking (in moderation) [Mean (Standard Deviation); unit: units on a scale] — How often have you and your parent talked about drinking in moderation is okay (Response categories 1=Never, 2=Occasionally, 3=Sometimes, 4= Often, 5 = Very often) Population: missing data explain differences in population analyzed
  units on a scale
    number analyzed (Participants) | 203 | 202 | 405
    (all) | 2.05 (1.36) | 2.08 (1.30) | 2.07 (1.33)
Overall communication about sex [Mean (Standard Deviation); unit: units on a scale] — Overall, how often you have talked to your parent about sex? (1=Never, 2=Occasionally, 3=Sometimes, 4=Often, 5= Very often) Population: 7 cases with missing data
  units on a scale
    number analyzed (Participants) | 203 | 201 | 404
    (all) | 2.65 (1.05) | 2.55 (1.11) | 2.60 (1.08)
Frequency for Topic Specific sexual activity [Mean (Standard Deviation); unit: units on a scale] — Average frequency created across 4 different sex topics (e.g., how being in a relationship might divert me from achieving my goals at school, how embarrassing it would be if I caught an STI -sexually transmitted infection) with higher scores indicating more topics discussed. Responses were reported on a likert type scale with 1= never, 2=occasionally, 3= sometimes, 4=often, and 5=very often. Scores ranged from 1 to 5. Population: one case missing data for variable
  units on a scale
    number analyzed (Participants) | 206 | 204 | 410
    (all) | 2.68 (1.06) | 2.62 (1.09) | 2.62 (1.09)
Communications regarding delaying sex [Mean (Standard Deviation); unit: units on a scale] — Communications regarding delaying sex based upon three questions with yes=1/no=0 responses summed: Have your parents told you that (i)you should not have sex, (ii)you should not be in a serious relationship while still in high school, (iii)you should not have sex because your religion or values forbid sex outside of marriage. Higher scores indicate more communications about delaying sex. Scores ranged from 0-3. Population: one case from each arm is missing data on this variable
  units on a scale
    number analyzed (Participants) | 205 | 204 | 409
    (all) | 1.23 (1.03) | 1.33 (1.10) | 1.28 (1.07)
Communication regarding health risks [Mean (Standard Deviation); unit: units on a scale] — Parent-teen communications score regarding health risks with sex were based upon two items: discussion that sex can result in pregnancy (y=1/n=0) and sex can result in sexually transmitted infections (y=1/n=0). Scores ranged from 0-2. Population: missing data for 4 cases
  units on a scale
    number analyzed (Participants) | 205 | 202 | 407
    (all) | 1.85 (0.46) | 1.81 (0.53) | 1.83 (0.50)
Number of Dating rules [Mean (Standard Deviation); unit: units on a scale] — Parental rules regarding dating were based upon 15 possible rules (parents must meet the date, check in once during the evening, parents must know destination, change plans-inform parent, address and phone number if going to party, no dates on school nights, no sex, no single dates, curfew, only go to agreed upon locations, use good judgment, be bentleman/lady, leave if uncomfortable, don't let someone domineer you, before sexually active discussion needed) with y=1/n=0 summed across the 15 items. Possible range 0-15. Population: 8 cases have missing data
  units on a scale
    number analyzed (Participants) | 201 | 202 | 403
    (all) | 11.19 (3.16) | 11.32 (3.10) | 11.26 (3.12)
Ever had sex [Count of Participants; unit: Participants] — Have you ever had sex (vaginal, oral, or anal)? (responses were yes=1/no=0) Population: Some teens did not answer the question
  Participants
    number analyzed (Participants) | 194 | 196 | 390
    (all) | 55 | 48 | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Teens Using Any Alcohol During Past 6 Months
Description: Have you had a drink of alcohol in the past 6 months? (A drink is a glass of wine, a can of beer, a wine cooler, a shot glass of liquor, or a mixed drink). (Response category yes=1/no=0). Range is 0-1. More frequent drinking is a worse outcome.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: Some teens were lost at follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Assigned Intervention, no Exposures: Assigned to intervention but had no exposure to alcohol component of the intervention.
- Control Condition: This group received information that was available on an NIAAA website
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposures | Control Condition
Number analyzed (Participants) | 99 | 101 | 201
Participants
  at 6 month follow-up: number analyzed (Participants) | 91 | 58 | 160
  at 6 month follow-up | 16 | 20 | 38
  at 12 month follow-up: number analyzed (Participants) | 87 | 57 | 162
  at 12 month follow-up | 14 | 23 | 43
  at 18 month follow-up: number analyzed (Participants) | 87 | 53 | 162
  at 18 month follow-up | 26 | 24 | 47
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposures vs Control Condition; 6 month follow-up. Among those assigned to intervention, dosage was assigned as 0 for no exposure, 1 for completing only the communication, and 2 for completing the alcohol component. A probit analysis predicting completion was conducted from baseline measures and an instrumental variable, inverse Mills' ratio (IMR) representing the underlying selection processes was included as a covariate accounting for factors related to program completion. All controls were assigned 0 dosage; Test type: Superiority; p < 0.01, Regression, Logistic; b=-.91, controlling for condition (experimental vs. control) , IMR, baseline measure of outcome variable, teen gender, age, & race; Odds Ratio (OR) = .40
Statistical Analysis 2: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposures vs Control Condition; 12 month follow-up. Among those assigned to intervention, dosage was assigned as 0 for no exposure, 1 for completing only the communication, and 2 for completing the alcohol component. A probit analysis predicting completion was conducted from baseline measures and an instrumental variable, inverse Mills' ratio (IMR) representing the underlying selection processes was included as a covariate accounting for factors related to program completion. All controls were assigned 0 dosage; Test type: Superiority; p < 0.10, Regression, Logistic; Odds Ratio (OR) = .58 — Controlling for condition (experimental vs. control) , IMR, baseline measure of outcome variable, teen gender, age, & race
Statistical Analysis 3: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposures vs Control Condition; 18 month follow-up. Among those assigned to intervention, dosage was assigned as 0 for no exposure, 1 for completing only the communication, and 2 for completing the alcohol component. All controls were assigned 0 dosage; Test type: Superiority; p = .077, Chi-squared; Chi-Square = 5.129

2. Primary Outcome: Frequency of Teen Alcohol Use Over Most Recent 30 Days Within Past 6 Months
Description: Over the past 30 days, how many times have you had a drink of alcohol? (response categories: 0=none, 1=once, 2=2-3 times, 3= once a week, 4=2-3 times a week. Range is 0-4.Higher score is more frequent drinking and a worse outcome.
Time Frame: Measured at 6, 12, & 18 months
Population: Missing responses and teens lost at follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Assigned Experimental, No Exposure: Assigned experimental, No exposure to alcohol component of intervention
Arm/Group | Smart Choices 4 Teens | Assigned Experimental, No Exposure | Control Condition
Number analyzed (Participants) | 97 | 100 | 201
units on a scale
  6 month follow-up: number analyzed (Participants) | 91 | 56 | 160
  6 month follow-up | .16 (.56) | .43 (.95) | .21 (.62)
  12 month follow-up: number analyzed (Participants) | 87 | 56 | 161
  12 month follow-up | .09 (.36) | .48 (.99) | .30 (.82)
  18 month follow-up: number analyzed (Participants) | 87 | 52 | 160
  18 month follow-up | .31 (.69) | .29 (.64) | .43 (.93)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Experimental, No Exposure vs Control Condition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Controled for condition (experimental vs. control) , IMR, baseline measure of outcome variable, teen gender, age, & race; b = -.47
Statistical Analysis 2: Comparison: Smart Choices 4 Teens vs Assigned Experimental, No Exposure vs Control Condition; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.01, Regression, Linear; Controlled for condition (experimental vs. control) , IMR, baseline measure of outcome variable, teen gender, age, & race; b = -.97
Statistical Analysis 3: Comparison: Smart Choices 4 Teens vs Assigned Experimental, No Exposure vs Control Condition; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p > 0.10, ANOVA; F = .85

3. Primary Outcome: Quantity of Alcohol Consumed by Teens on Drinking Days for the Most Recent 30 Days Within the Past Six Months
Description: Over the past 30 days, how many drinks did you usually have on days you drank? (response categories: 0= less than one, 1, 2, 3, 4, 5, 6, 7= more than six). Range is 0-7. Higher scores represent more drinking and worse outcome.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: Cases lost to follow-up and for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smart Choices 4 Teens | Assigned Experimental, No Exposure | Control Condition
Number analyzed (Participants) | 97 | 100 | 201
units on a scale
  6 month follow-up: number analyzed (Participants) | 91 | 56 | 160
  6 month follow-up | .16 (.64) | .46 (1.22) | .32 (1.13)
  12 month follow-up: number analyzed (Participants) | 87 | 56 | 161
  12 month follow-up | .13 (.64) | .61 (1.28) | .40 (1.13)
  18 month follow-up: number analyzed (Participants) | 88 | 100 | 201
  18 month follow-up | .46 (1.18) | .45 (1.26) | .60 (1.48)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Experimental, No Exposure vs Control Condition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.10, Regression, Linear; b = -.22 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Smart Choices 4 Teens vs Assigned Experimental, No Exposure vs Control Condition; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, Regression, Linear; b = -.24 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Smart Choices 4 Teens vs Assigned Experimental, No Exposure vs Control Condition; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p > 0.10, ANOVA; F = 0.43

4. Primary Outcome: Count of Teens Who Were Drunk or Very, Very High During the Past 6 Months
Description: Over the past 6 months, how many times have you gotten drunk or very, very high on alcohol? (Response categories: 0=none, 1=once a month, 2=2-3 times a month, 3=once a week, 4= 2-3 times a week, 5=daily or almost daily). Range is 0-5. Higher score represents more drunkenness and a worse outcome.
Time Frame: Measured at 6, 12, & 18 months
Population: Within the experimental group, 49.5% completed the alcohol component of the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Assigned Experimental, no Exposure: This group had no exposure to the intervention relating to sexual communication and behaviors
Arm/Group | Smart Choices 4 Teens | Assigned Experimental, no Exposure | Control Condition
Number analyzed (Participants) | 99 | 100 | 201
score on a scale
  6 month follow-up: number analyzed (Participants) | 91 | 57 | 160
  6 month follow-up | .10 (.40) | .26 (.96) | .23 (.91)
  12 month follow-up: number analyzed (Participants) | 87 | 55 | 162
  12 month follow-up | .08 (.35) | .44 (1.46) | .39 (1.20)
  18 month follow-up: number analyzed (Participants) | 87 | 53 | 161
  18 month follow-up | .21 (.61) | .26 (1.00) | .45 (1.30)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Experimental, no Exposure vs Control Condition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .10, Regression, Linear; [statistical method as in outcome 2, analysis 2]; b = -.16
Statistical Analysis 2: Comparison: Smart Choices 4 Teens vs Assigned Experimental, no Exposure vs Control Condition; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, Regression, Linear; [statistical method as in outcome 2, analysis 2]; b = -.26
Statistical Analysis 3: Comparison: Smart Choices 4 Teens vs Assigned Experimental, no Exposure vs Control Condition; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p > 0.10, ANOVA; F = 1.550

5. Primary Outcome: Frequency of Parental Approval for Teen Drinking (in Moderation)
Description: How often have you and your parent talked about drinking in moderation is okay (Response categories 1=Never, 2=Occasionally, 3=Sometimes, 4= Often, 5 = Very often). Range is 1-5 and higher scores means more parental approval of teen drinking and is a worse outcome.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: Across time, there was loss of sample at follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposures | Control Condition
Number analyzed (Participants) | 101 | 101 | 203
units on a scale
  6 month follow-up: number analyzed (Participants) | 90 | 58 | 203
  6 month follow-up | 1.99 (1.31) | 2.59 (1.40) | 2.26 (1.35)
  12 month follow-up: number analyzed (Participants) | 88 | 56 | 162
  12 month follow-up | 2.16 (1.29) | 2.66 (1.55) | 2.19 (1.27)
  18 month follow-up: number analyzed (Participants) | 89 | 53 | 161
  18 month follow-up | 2.12 (1.40) | 2.57 (1.31) | 2.13 (1.28)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposures vs Control Condition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, Regression, Linear; b = -.35 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposures vs Control Condition; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p > 0.10, Regression, Linear; b = -.02 — [estimate comment as in outcome 1, analysis 2]

6. Primary Outcome: Frequency of Teen- Parent Communications Regarding Sex
Description: Overall, how often you have talked to your parent about sex? (1=Never, 2=Occasionally, 3=Sometimes, 4=Often, 5= Very often). Range 1-5. Higher scores represent a better outcome.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: The rows represent 3 different follow-up periods and the number of cases analyzed varied because the responses at follow-up varied.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Assigned Intervention, no Exposure: This group was assigned to the intervention but had no exposure to the relationship component of the intervention.
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposure | Control Condition
Number analyzed (Participants) | 81 | 67 | 165
score on a scale
  6 month follow | 2.46 (0.99) | 2.18 (1.28) | 2.19 (1.20)
  12 month follow up: number analyzed (Participants) | 76 | 66 | 163
  12 month follow up | 2.45 (1.17) | 2.02 (1.09) | 2.23 (1.16)
  18 month follow-up: number analyzed (Participants) | 78 | 63 | 161
  18 month follow-up | 2.46 (1.17) | 1.97 (1.08) | 2.07 (1.04)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposure vs Control Condition; Among those assigned to intervention, dosage was assigned as 0 for no exposure, 1 for completing some of the program, and 2 for completing the relationship component. A probit analysis predicting completion was conducted from baseline measures and an instrumental variable, inverse Mills' ratio (IMR) representing the underlying selection processes was included as a covariate accounting for factors related to program completion. All controls were assigned 0 dosage; Test type: Superiority; p < 0.01, generalized estimating equations; b = .299 — [estimate comment as in outcome 1, analysis 2]

7. Primary Outcome: Frequency of Teen-parent Communications About Specific Sexual Topics
Description: Average frequency created across 4 different sex topics (i. how being in a relationship might divert me from achieving my goals at school, ii. how embarrassing it would be if I caught an STI -sexually transmitted infection, iii. sexual relationships can impact health, iv. how pregnancy would be embarassing) with responses being never=1, occasionally=2, sometimes=3, often=4, very often=5 for a full range of 1-5. Across the 4 different sex topics the sums ranged from 4-20 and average was created by dividing the score by 4, with higher scores indicating more both topics and higher frequency of discussions taking place for a final full range of 1-5.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: The number analyzed varies across rows because the rows represent different follow-up periods and participation varied across follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposure | Control Condition
Number analyzed (Participants) | 82 | 67 | 164
score on a scale
  Frequency of sexual communication at 6 month follow-up: number analyzed (Participants) | 82 | 67 | 162
  Frequency of sexual communication at 6 month follow-up | 2.60 (1.11) | 2.23 (1.06) | 2.27 (1.10)
  Frequency of sexual communication at 12 month follow-up: number analyzed (Participants) | 79 | 67 | 164
  Frequency of sexual communication at 12 month follow-up | 2.50 (1.12) | 2.03 (0.93) | 2.36 (1.11)
  Frequency of sexual communication at 18 month follow-up: number analyzed (Participants) | 80 | 63 | 164
  Frequency of sexual communication at 18 month follow-up | 2.47 (1.10) | 2.50 (1.12) | 2.23 (1.06)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposure vs Control Condition; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < .03, generalized estimating equations; b = .268

8. Primary Outcome: Count of Teen-parent Communications Regarding Delaying Sexual Activity
Description: Communications regarding delaying sex based upon three questions with yes=1/no=0 responses summed: Have your parents told you that (i)you should not have sex, (ii)you should not be in a serious relationship while still in high school, (iii)you should not have sex because your religion or values forbid sex outside of marriage. Higher scores indicate more communications about delaying sex. Range is 0-3. Higher scores represent a better outcome.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: The three rows represent different follow-up periods and there are different response rates across follow-up periods.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposure | Control Condition
Number analyzed (Participants) | 82 | 66 | 164
score on a scale
  Communication regarding delay sex at 6 month follow-up: number analyzed (Participants) | 82 | 66 | 159
  Communication regarding delay sex at 6 month follow-up | 1.13 (1.09) | 0.85 (0.98) | 0.98 (1.04)
  Communication regarding delay sex at 12 month follow-up: number analyzed (Participants) | 78 | 65 | 164
  Communication regarding delay sex at 12 month follow-up | 1.09 (1.11) | 1.02 (1.08) | 1.07 (1.10)
  Communication regarding delay sex at 18 month follow-up: number analyzed (Participants) | 80 | 63 | 161
  Communication regarding delay sex at 18 month follow-up | 0.98 (1.04) | 0.75 (1.00) | 0.95 (1.11)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposure vs Control Condition; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p > 0.10, generalized estimating equations; b = .075 — [estimate comment as in outcome 1, analysis 2]

9. Primary Outcome: Count of Teen-parent Communications Regarding Health Risks Associated With Sex
Description: Parent-teen communications score regarding health risks with sex were based upon two items: discussion that sex can result in pregnancy (y=1/n=0) and sex can result in sexually transmitted infections (y=1/n=0). Range is 0-2. Higher scores represent a better outcome.
Time Frame: Past 6, 12, & 18 months
Population: Each row represents a different follow-up time period and the number of respondents varied across the time periods.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposure | Control Condition
Number analyzed (Participants) | 88 | 65 | 164
score on a scale
  Communications on Health Risks at 6 month follow-up: number analyzed (Participants) | 82 | 65 | 158
  Communications on Health Risks at 6 month follow-up | 1.63 (0.71) | 1.35 (0.89) | 1.51 (.77)
  Communications on Health Risks at 12 month Follow-up | 1.53 (0.77) | 1.40 (0.86) | 1.54 (0.79)
  Communications on Health Risk at 18 month follow-up: number analyzed (Participants) | 88 | 63 | 162
  Communications on Health Risk at 18 month follow-up | 1.49 (0.83) | 1.27 (0.90) | 1.38 (0.86)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposure vs Control Condition; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p > 0.10, generalized estimating equations; b = 0.051 — [estimate comment as in outcome 1, analysis 2]

10. Primary Outcome: Count of Parental Dating Rules
Description: Parental rules regarding dating were based upon summing the yes (=1) response to 15 possible rules: parents must meet date, check in/call during date, parents must know destination, parents must know change of plans, address and phone number needed for parties, no dates on school nights, no sex, no sigle dates, curfew, only agreed upon locations, use good judgment, be gentleman/lady, leave if uncomfortable (y=1/n=0). Range is 0-15. Higher scores represent better outcomes.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: There are 3 follow-up periods and the numbers analyzed vary across these follow-up periods
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Condition: This group was provided with websites where information was available regarding ...
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposure | Control Condition
Number analyzed (Participants) | 82 | 65 | 163
score on a scale
  Dating Rules-Teen report 6 month follow-up | 11.48 (2.97) | 10.18 (3.91) | 10.77 (3.57)
  Dating rules, teen report, 12 month follow-up: number analyzed (Participants) | 77 | 65 | 162
  Dating rules, teen report, 12 month follow-up | 11.04 (3.47) | 10.42 (3.57) | 10.72 (3.44)
  Dating rules, teen report, 18 month follow-up: number analyzed (Participants) | 78 | 62 | 160
  Dating rules, teen report, 18 month follow-up | 11.01 (3.29) | 9.53 (3.59) | 10.08 (4.09)
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposure vs Control Condition; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.05, generalized estimating equations; b = 0.72

11. Primary Outcome: Count of Teens Who Have Ever Had Sex Over Their Lifetime
Description: Have you ever had sex (vaginal, oral, or anal)? (responses were yes=1/no=0). Range was 0-1. Higher score is worse outcome risk.
Time Frame: Measured at baseline, 6, 12, & 18 months
Population: The three rows reflect different follow-up periods, teens were lost to follow-up in subsequent waves
Measure: Count of Participants; unit: Participants
Arm/Group | Smart Choices 4 Teens | Assigned Intervention, no Exposure | Control Condition
Number analyzed (Participants) | 60 | 50 | 122
Participants
  ever had sex at 6 month follow-up | 17 | 15 | 37
  ever had sex at 12 month follow-up: number analyzed (Participants) | 59 | 47 | 117
  ever had sex at 12 month follow-up | 17 | 20 | 39
  ever had sex at 18 month follow-up: number analyzed (Participants) | 58 | 39 | 111
  ever had sex at 18 month follow-up | 19 | 21 | 46
Statistical Analysis 1: Comparison: Smart Choices 4 Teens vs Assigned Intervention, no Exposure vs Control Condition; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p > 0.10, Chi-squared

ADVERSE EVENTS:
Time Frame: Over three years of the study
Description: None of the parents or teens were exposed to any experimental condition that threatened life. There was not physical or medical intervention. This was a prevention program that was designed to address behavioral health issues.
Arm/Group | Smart Choices 4 Teens | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/205
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/205
Other Adverse Events (participants affected / at risk) | 0/206 | 0/205

LIMITATIONS AND CAVEATS:
This sample was drawn from a nationwide sample of families compiled by panel vendors. Smart Choices 4 Teens is family-based, designed to promote healthy choices by teens related to alcohol use and relationships. It is not a treatment program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT03521115/Prot_SAP_000.pdf